CLINICAL TRIAL: NCT04192890
Title: Efficacy and Safety Assessment of Nanoknife (AngyoDynamics, USA) for Irreversible Electroporation (IRE) of Localized Prostate Cancer
Brief Title: Efficacy and Safety Assessment of IRE of Localized Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sechenov-IRE19
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate; Irreversible Electroporation; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IRE patients (Experimental): patients who will underwent 'Focal irreversible electroporation of the prostate cancer'
  Interventions: Device: Focal irreversible electroporation of the prostate cancer

INTERVENTIONS:
Device: Focal irreversible electroporation of the prostate cancer — Irreversible electroporation is a non-thermal tissue ablation technique in which short duration electrical fields are used to permanently permeabilize the cell membrane.

SUMMARY:
The purpose of this study is to evaluate safety and short-term oncological efficacy of the NanoKnife Irreversible Electroporation System for localised prostate cancer.

Irreversible electroporation (IRE) is the method of focal treatment for prostate cancer, which is already proven by FDA as method of the surgical ablation of soft tissue. It has not received clearance for the therapy or treatment of any specific disease or condition.

DETAILED DESCRIPTION:
Detailed Description:

Irreversible electroporation is a newly developed non-thermal tissue ablation technique in which short duration electrical fields are used to form permanent nanoscale defects in the cell membrane which leads to cell apoptosis. Thus, IRE is a non-thermal technique, which means that changes associated with tissue freezing or heating are not relevant.

Moreover, animal studies of IRE in the canine prostate have demonstrated that structures such as ejaculatory ducts, neurovascular bundles, blood vessels, and the urethra heal normally after ablation. The reason is that collagen matrix during treatment with IRE is not destroyed thus allowing for a large structures (blood vessels, nerves, etc.) to heal normally.

This study is a prospective and non-randomized with one group of 12 patients eligible for focal therapy of prostate cancer with IRE (eligibility defined by this protocol).

Before the surgery all patients will underwent transperineal MRI-fusion biopsy to localize the prostate cancer foci.

Objectives of the study: to asses safety of IRE in patients with localized PCa, to asses short-term oncologic efficacy of IRE in patients with localized PCa, to asses functional outcomes after IRE.

All patients will be followed up for 1 year (each 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Verified with MR-fusion biopsy localized Pca
* PSA < 20 ng/ml
* Gleason score 3+3=6; 3+4=7 OR Grade Group 1 and 2
* Life expectancy > 10 years
* No post-void residual urine or infravesical obstruction

Exclusion Criteria:

* patients with artificial cardiac pacemaker
* patients not eligible for general anesthesia
* patients after primary Pca treatment
* hormonal therapy six months before the study
* radiotherapy of pelvic organs
* urinary infection
* extracapsular Pca
* patients with metastatic lesions

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Presence of the prostate
Enrollment: 12 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
PSA level | 3 months, 6 months, 9 months, 12 months
  Stable decrease of PSA level after surgery (<1 ng/ml)
Complications | 1 year
  Short and long term surgical complications according to Clavien-Dindo

SECONDARY OUTCOMES:
IPSS (International Prostate Symptom Score, range from 5 to 30 | 1 year
  International Prostate Symptom Score
QoL (Quality of Life score, range 1-6) | 1 year
  Quality of Life Score
Qmax | 1 year
  Maximal urine flow rate
IIEF | 1 year
  International Index of Erectile Function - Erectile function assessment (range 1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided